CLINICAL TRIAL: NCT02861690
Title: Phase II Study of Liposomal Paclitaxel With Nedaplatin as First-line in Advanced or Recurrent Esophageal Carcinoma
Brief Title: Liposomal Paclitaxel Combined Nedaplatin in Treatment of Advanced or Recurrent Esophageal Carcinoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Ruihua Xu, professor, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Esophageal cancer 001
Record Dates: First submitted 2016-07-28; First posted 2016-08-10 (Estimated); Last update posted 2016-08-10 (Estimated); Status verified 2016-08

CONDITIONS: Esophageal Carcinoma
Keywords: Esophageal Cancer; nedaplatin; Liposomal Paclitaxel
MeSH Terms: conditions — Esophageal Neoplasms | interventions — nedaplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment group (Experimental): patients received Liposomal Paclitaxel and Nedaplatin every 21 days until the presence of progressive disease or unacceptable toxicity
  Interventions: Drug: Liposomal Paclitaxel; Drug: Nedaplatin

INTERVENTIONS:
Drug: Liposomal Paclitaxel — Patients received Liposomal Paclitaxel 175mg/m2 every 21 days until the presence of progressive disease or unacceptable toxicity.
Drug: Nedaplatin — Patients received Nedaplatin80mg/m2 every 21 days until the presence of progressive disease or unacceptable toxicity.

SUMMARY:
The purpose of this study is to evaluate the safety, tolerance and efficacy of Liposomal Paclitaxel With Nedaplatin as First-line in patients with Advanced or Recurrent Esophageal Carcinoma

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the safety, tolerance and efficacy of Liposomal Paclitaxel With Nedaplatin as First-line in patients with Advanced or Recurrent Esophageal Carcinoma.Patients receive Liposomal Paclitaxel 175mg/m2 and Nedaplatin 80mg/m2 every 21 days until the presence of progressive disease or unacceptable toxicity.

ELIGIBILITY:
Inclusion Criteria:

Inclusion Criteria:

1. histological confirmed advanced metastatic or recurrent esophageal cancer
2. age between 18 and 80 years
3. ECOG performance status of 0 to 2
4. life expectancy ≥ 12 weeks
5. has evaluable disease by Response Evaluation Criteria in Solid Tumors (RECIST)
6. at least one prior chemotherapy regimen
7. adequate bone marrow function as defined by absolute neutrophil count more than or equal to 2000/mm3
8. platelet count more than or equal to 100,000/mm3 and hemoglobin more than or equal to 8 g/dL
9. adequate renal function defined by creatinine less than or equal to 1.25 × upper limit of normal(ULN) and creatinine clearance more than or equal to 60mL/min,
10. adequate liver function defined by bilirubin less than or equal to 1.0×ULN aspartate transferase(AST) and alanine transferase(ALT) less than or equal to 2.5 ×ULN.

Exclusion Criteria:

1. other primary malignancy
2. symptomatic central nervous system metastasis
3. pregnancy or lactation
4. cardiovascular events such as myocardial infarction in the previous 6 months or congestive heart failure
5. ongoing infection

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2010-01; Primary Completion 2015-09 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Response rate | from date of baseline measured to date of first CT evaluation，Up to 3 months
  To assess the response rate of Liposomal Paclitaxel and Nedaplatin in patients with pretreated advanced or recurrent esophageal carcinoma. Possible evaluations include: Complete Response (CR): Disappearance of all target lesions. Partial Response (PR): At least a 30% decrease in the size of target lesions. Progressive Disease (PD): At least a 20% increase in the size of target lesions. Stable Disease (SD): Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD.

SECONDARY OUTCOMES:
progression-free survival | from date of baseline to the date of first documented progression or date of death from any cause, whichever came first, assessed up to 24 months
  Progression-free survival (PFS) is defined as the time from the date of study enrollment to the date of objectively determined PD or death from any cause, whichever comes first. For patients who are still alive at the time of analysis, and who do not have PD, PFS will be censored at the date of the last objective progression-free disease assessment.
overall survival | baseline to date of death from any cause，up to 2 approximately years
  Overall survival is defined as the time from the date of study enrollment to the date of death from any cause.
Number of Participants With Adverse Events (Toxicity) | Up to 30 days post last dose
  Number of participants with treatment-related adverse events as assessed by CTCAE.

CONTACTS AND LOCATIONS:
Overall Officials: Rui-hua Xu, Study Chair — Sun Yat-sen UniversityCancer center
Locations (1):
- Medical Oncology,Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No